CLINICAL TRIAL: NCT06259201
Title: Vagus Nerve Stimulation for Autonomic Dysregulation in Individuals With Developmental Disorders
Brief Title: Vagus Nerve Stimulator for Autism and Other Developmental Disorders
Acronym: VNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Institute for Basic Research (Other Government)
Collaborators: Boston Children's Hospital (Other); Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYInstitute
Record Dates: First submitted 2023-07-07; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder; Intellectual Disability; Autonomic Nervous System; Developmental Disability
Keywords: Vagus Nerve Stimulation
MeSH Terms: conditions — Autism Spectrum Disorder; Intellectual Disability; Developmental Disabilities | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Each participant will begin the study with the first baseline phase (1 month).
  Each participant will receive 1 month of VNS administered twice per day (AM & PM).
  During the study, the participant (or legal guardian) and the study team can decide whether to:
  1. Complete 1 month of VNS and go to Baseline 2 (ABA design); or
  2. Continue with 2 months of VNS and go to Baseline 2 (ABBA design); or
  3. Continue with 3 months of VNS and go to Baseline 2 (ABBBA design)
  Each participant will have 1-month, 3-month, and 6-month follow-ups with the study team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Vagus Nerve Stimulation (VNS) (Experimental): Single-subject design: ABA, ABBA, or ABBBA
  This study allows for a flexibility in the duration of research participation depending on one's response. The participant will be able to select one of the three design options (1, 2, or 3 months of VNS twice per day) in consultation with the study staff. That is, after the initial 1-month trial of VNS, the participant may choose to extend the VNS two more times (i.e., 1 or 2 months), for a total of 90 days.
  Interventions: Device: Vagus Nerve Stimulation

INTERVENTIONS:
Device: Vagus Nerve Stimulation — Vagal nerve stimulation (VNS) involves the use of a device to stimulate the vagus nerve with electrical impulses twice per day (AM & PM) for two minutes each. It is an approved treatment for treatment resistant epilepsy and depression.
  Other Names: gammaCore

SUMMARY:
The goal of this flexible single-subject design vagus nerve stimulation (VNS) study is to examine the behavioral, cognitive, and biorhythmic effects of VNS in children and adults with autism and developmental disabilities. The main aims are:

* Pilot the creation of a profile for those who will respond to VNS with the long-term goal of designing clinical trials.
* Examine the effects of VNS on a broad range of symptoms.

Participants will select between 1, 2, or 3 months of daily VNS treatment and complete study visits each month.

DETAILED DESCRIPTION:
Intellectual and developmental disabilities (IDD) cover a wide variety of disorders. Although we know the causes of some of the disorders and some of them could even be prevented (e.g., lead exposure), most causes remain unknown. Without having a clear understanding of the causes, prevention is very difficult to achieve. Previous studies have shown abnormal autonomic nervous system (ANS) regulations in young children with autism spectrum disorder (ASD) and these abnormalities are also observed during sleep. ANS is the part of the nervous system that controls the unconscious bodily functions, such as breathing, heart beating, and digestion.

The vagus nerve strongly influences these autonomic functions including digestion, breathing, heart rate variability, and metabolic function and central nervous system (CNS) activity that affect mood, pain, stress management, sleep, and even memory and cognitive functions. The vagal influence over neurotransmitter release has been implicated in the regulation of inflammation and immune cell activity.

Here, we are using a non-invasive vagus nerve stimulator to monitor changes in cognitive function and other symptoms in people with IDD, both with and without ASD. The device is FDA-approved for migraine and cluster headaches in people 12 years and older. VNS activates the vagus nerve with mild electrical stimulation through the skin.

Rather than embarking on a rigorously designed study, we will conduct a series of single-subject studies that reflects each participant's symptoms. We will select the most appropriate dependent variables based on each person's symptom presentation.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adults aged 12-40 with intellectual and developmental disability (IDD) and/or autism spectrum disorder (ASD). Participants who are decisionally-impaired will be eligible with assent.
2. Able to tolerate wearing an Apple Watch, EEG, and sit for a neurocognitive test
3. Be on a stable dose of psychotropic medication for at least one month prior to enrollment
4. Agree not to initiate new or change existing medications or behavior intervention

Exclusion Criteria:

1. Have an active implantable medical device (e.g., pacemaker, implanted hearing aid, etc.) or a metallic device, such as a stent, bone plate, or bone screw
2. Have a comorbid physical or psychiatric disorder which would disrupt ability to tolerate vagal stimulation or comply with study demands (e.g., insulin dependent diabetes, bipolar, etc.)
3. Vagus nerve lesion, damage, or structural abnormality (e.g., lymphadenopathy, neoplasm, previous surgery), or pain (e.g., dysesthesia, neuralgia and/or cervicalgia)
4. Current or past history of neurological disorders or trauma, including uncontrolled epilepsy and head injury.
5. Current or recent (within 12 months) participation in a clinical trial of a drug or a medical device.
6. Use of drugs (within 4 weeks) that affect the autonomic nervous system (beta blockers, beta stimulant, etc.).
7. Use of marijuana (including medical marijuana) for any indication
8. Any condition per the investigators' clinical judgment that precludes participation in the study (e.g., pregnancy).
9. Lack of capacity to consent and without a legally authorized representative (LAR) who is a parent, spouse, or an adult child.
10. Living in a residential program (e.g., group home)
11. Wards of state

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-Community (ABC-C) | Change measured once per month for 3, 4, or 5 months
  The ABC-C is a 58-item questionnaire consisting of five subscales: Irritability, Lethargy, Inappropriate Speech, Hyperactivity, and Stereotypy. Minimum score = 0, maximum score = 174. Higher scores indicate more severity.
Pervasive Developmental Disorder Behavior Inventory (PDDBI) | Change measured once per month for 3, 4, or 5 months
  The PDDBI is an informant-based assessment that examines treatment effectiveness and differentiates ASD from other conditions. It consists of the following Approach/Withdrawal Problems: 1) Sensory/Perceptual Approach, 2) Ritualisms/Resistance to Change, 3) Social Pragmatic, 4) Semantic Pragmatic, 5) Arousal Regulation, 6) Specific Fears, 7) Aggressiveness. Under Receptive/ Expressive Social Communication Abilities, there are 1) Social Approach Behaviors, 2) Expressive Language, and 3) Learning, Memory, and Receptive Language. Higher T scores on Approach/Withdrawal Problems indicate more symptom severity and higher T scores on Receptive/Expressive Social Communication indicate more skills.
Behavior Rating Inventory of Executive Function (BRIEF) | Change measured once per month for 3, 4, or 5 months
  The BRIEF is an informant-based assessment that contains 63 (preschool age) 86 (school age) items with eight subdomains of executive function: 1) Inhibit, 2) Shift, and 3) Emotional Control subdomains together result in an additional composite Behavioral Regulation Index. The subdomains 4) Initiate, 5) Working Memory, 6) Plan/Organize, 7) Organization of Materials, and 8) Monitor provide a composite Metacognition Index. The indexes are also combined to obtain an overall Global Executive Composite. Higher T scores indicate more symptom severity.
The Symptom Checklist-90-Revised (SCL-90-R) | Change measured once per month for 3, 4, or 5 months
  The SCL-90-R is a questionnaire designed to evaluate a broad range of psychological problems and symptoms of psychopathology. It is also useful in measuring treatment outcomes. Higher T scores indicate more symptom severity.
Repetitive Behavior Scale-Revised (RBS-R) | Change measured once per month for 3, 4, or 5 months
  The RBS-R is a 44-item questionnaire that is used to measure the breadth of repetitive behavior in people with ASD. The RBS-R consists of six subscales including: Stereotyped, Self-injurious, Compulsive, Routine, Sameness, and Restricted Behaviors. Minimum score = 0; maximum score = 136. Higher scores indicate more severity.
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) (Y-BOCS) | Change measured once per month for 3, 4, or 5 months
  The Y-BOCS is a measurement tool for OCD. It is not a diagnostic tool. Rather, it is a scale used to gauge the severity and nature of OCD symptoms and to monitor improvement. Higher scores indicate severity. Minimum score = 0; maximum score = 40. Higher scores indicate more severity.

SECONDARY OUTCOMES:
Neurocognitive assessment | Change measured once per month for 3, 4, or 5 months
  An online tablet-based nonverbal (i.e., visually presented on an iPad) neurocognitive tasks to examine specific components of cognition, particularly those associated with executive function skills related to frontal and medial temporal regions of the brain (e.g., planning, episodic memory, processing speed) will be collected. Subtests are specifically selected for IDD/ASD and graded in difficulty, minimizing floor and ceiling effects.
Electro-encephalogram (EEG) | Change measured once per month for 3, 4, or 5 months
  EEG is a non-invasive test that records electrical activity in the brain. It works by picking up brain waves via electrodes that are attached to the scalp. EEG data will be collected for 10-15 mins while the participant is awake.
  Power, sample entropy, Lyapunov exponent, detrended fluctuation analysis, correlation dimension, and recurrence quantitative analysis (RQA) values on all frequency bands (delta, theta, alpha, beta, gamma, and gamma+) will be computed using a portable headset.
Biorhythmic motion measurements | Change measured once per month for 3, 4, or 5 months
  On-body sensors: Patterns of motor and heart variability in the form of time series collected to align the signals for before, during, and after VNS comparison.
  OFF-body sensors: Time series of digital data to extract patterns of variability and stochastic signatures aligned to the stimulation.

OTHER OUTCOMES:
Non-verbal Pain Measure | Twice per day for 3, 4, or 5 months
  Non-verbal Pain and Discomfort Indicators for those participants who are non-verbal. Minimum score = 0; maximum score = 8. Higher scores indicate more pain and discomfort.
Columbia-Suicide Severity Rating Scale (C-SSRS) | every 4 weeks for 3, 4, or 5 months
  C-SSRS is a suicidal ideation and behavior rating scale to evaluate suicide risk. It rates one's degree of suicidal ideation on a scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent and behaviors." An answer of "yes" to any of the six questions may indicate a need for referral and an answer of "yes" to questions 4, 5 or 6 indicate high-risk.
Clinical Global Impression Scale Severity & Improvement (CGI-S, CGI-I) | Change measured once per month for 3, 4, or 5 months
  measures of symptom severity, treatment response and the efficacy of treatments. Minimum score = 1; maximum score = 7. Higher scores indicate more severity (CGI-S) or worsening (CGI-I).

CONTACTS AND LOCATIONS:
Overall Officials: Helen Yoo, Ph.D., Principal Investigator — New York State Institute for Basic Research
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, New York, New York
  - New York State Institute for Basic Research, Staten Island, New York

IPD SHARING:
Plan to Share IPD: No